CLINICAL TRIAL: NCT06211621
Title: Admission Pattern Among Children With Gastro-intestinal Infections Before and During the Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Region Zealand (Other)
Responsible Party: Principal Investigator, Maren Rytter, Consultant, PhD, clinical associate professor, Region Zealand
Other Study IDs: R-21041034
Record Dates: First submitted 2023-12-29; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Gastroenteritis; Rota Virus Gastroenteritis; Dehydration in Children; Infectious Disease; COVID-19 Pandemic; Norovirus Infections
Keywords: gastroenteritis; indirect effects; lockdown; epidemic; pandemic; children; Denmark; dehydration; diarrhea
MeSH Terms: conditions — Gastroenteritis; Communicable Diseases; COVID-19; Caliciviridae Infections; Dehydration; Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During the Covid-19 pandemic, admission patterns for infections other than Covid-19 have changed dramatically among children worldwide.

Particularly admissions due to respiratory infections and later invasive streptococcal infections have been well documented.

However, few studies have compared rates af gastro-intestinal infections during the pandemic with the previous years.

This study aims to compare the number and characteristics of children hospitalized with gastrointestinal infections before the COVID-19 pandemic, to the first strict lockdown in 2020 and to the second, less strict lockdown in 2021.

A retrospective review of medical records will be performed, of patients aged 1 month to 5 years admitted with gastroenteritis at the pediatric department at Slagelse Hospital in Denmark over a period from 2017 to 2021.

DETAILED DESCRIPTION:
Admission patterns among children with non-Covid gastro-intestinal infections before and during the Covid-19 pandemic

1. Purpose To compare incidence of and clinical characteristics of children admitted with gastro-intestinal infections during the Covid-19 pandemic relative to prepandemic seasons.

This will improve understanding of the indirect effects of the Covid-19 pandemic

HYPOTESES

1. During the winter-spring months after the lock-down in 2020 fewer children were admitted with gastro-intestinal infections, relative to the winter-spring months of the pre-pandemic years, while more children were admitted during the winter-spring season of 2021 relative to pre-pandemic years.
2. Children admitted during the winter-spring season of 2021 were more severely ill, and older than children admitted during the prepandemic seasons.

2. BACKGROUND During the COVID-19 pandemic, admission patterns for infections other than Covid-19 have changed dramatically among children worldwide. [1][2]

During the first lockdown of 2020 a dramatic decline in children admitted with infections other than Covid-19 was reported worldwide. [1] Initially, concerns was expressed that this decline could be due to fear of seeking health care, or other barriers to access health care. For example, children with newly diagnosed diabetes in Germany were reported to present with ketoacidosis more frequently than before the pandemic. [3] [4] However, the main reason is likely to be reduced social contact limiting the spread of many other infections.

Later, reports of delayed epidemics - for example, the expected annual epidemic of respiratory syncytial virus did not occur in the winter of 2021, only to occur later and unexpectedly in the summer. This was first reported in Australia, and later in the Northern hemisphere, including Denmark [5][6].

Particularly admissions due to respiratory infections and later invasive streptococcal infections have been well documented.

Annual epidemics of viral gastrointestinal infections are known to occur in children in the winter and spring months, most caused by rotavirus infections. In the spring of 2021 many Danish paediatricians experienced an unusual surge of children admitted with gastroenteritis, and the general impressioin was that children werre older and more severely dehydrated than during previous seasons.

However, it has not yet been assessed whether gastroenteritis rates were indeed higher in 2021 during the pandemic, compared to the previous years, and whether the admitted children differed from children admitted before the pandemic.

Accordingly, this is what is planned to investigate with the current project.

Hopefully, the project may improve understanding of how well-known and regular epidemics are affected indirectly by the emergence of new diseases - and by the public health measures applied to prevent its spread. This may potentially inform management of future pandemics to reduce the harms, directly as well as indirectly.

3. METHODS Study design

Retrospective review of patient files among children admitted with gastrointestinal infections in the paediatric department of Slagelse Hospital, during the spring-winter months (january to june) of three periods:

* pre-pandemic: january - june of 2017, 2018 and 2019 as well as january and february of 2020
* early pandemic: march-june 2020
* late pandemic: january - june of 2021

Participants:

Children aged from >1 months to <5 years with symptoms of gastroenteritis admitted to the paediatric department in Slagelse Hospital

Patient files will be identified in the electronic health record (EPIC) by a search of diagnoses such as "gastroenteritis", "rotavirus", "vomiting", "diarrhea", "dehydration". Each patient file will be evaluated by a doctor, and the child will be included if it is confirmed that the child was admitted with symptoms of gastrointestinal infection.

Data From the identified patient files anonymized data will be retrieved on age, gender, preexisting disease, past history, family type, breastfeeding, nutritional status, estimated degree of dehydration, as well as symptoms and clinical findings on admission, treatment given, duration of admission as well as microbiology and biochemical data.

Handling of data Data will be handles according to GDPR regulations. Anonymized data will be entered into a secured database (RedCAP) and analysed using the statistical package Stata.

5. Funding The Slagelse hospitals research fund has funded three months of salary for a junior doctor and a medical student to type data and conduct the study

6. Ethical issues and authorisation: The project has been registered on the research directory of Region Zealand (Regions Sjællands Interne Forskningsfortegnelse, no. REG-087-2021.)

The committee of research ethics of Region Zealand has stated that the study does not need reaserch ethical approval according to Danish Law, as it only involves retrieval of data from hospital files.

Regions Zealand has approved that anonymized data is collected from patient files without consent from the parents (Ref nr: R-21041034)

7. PUBLICATION OF RESULTS The results of the project (whether positive, negative or inconclusive) will be submitted for publication to a peer reviewed scientific journal.

ELIGIBILITY:
Inclusion Criteria:

* Children admitted to Slagelse hospital
* aged >1 month and <5 years
* symptoms of gastrointestinal infection
* admitted during the months of january-june of 2017, 2018, 2019, 2020 and 2020

Exclusion Criteria:

none

Ages: 1 Month to 59 Months | Sex: All
Age Groups: Child
Study Population: Children aged >1 month and <5 years admitted with symptoms of gastroenteritis at Slagelse Hospital during the months of january-june of 2017, 2018, 2019, 2020 and 2020
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
incidence of admission with gastroeneteritis in children | five years (2017 to 2021)
  number of children admitted/1000 children per month

SECONDARY OUTCOMES:
age of children admitted | five years (2017 to 2021)
  age in month
severity of illness | five years (2017 to 2021)
  proportion treated with IV fluids, base excess in blood, duration of admission

CONTACTS AND LOCATIONS:
Overall Officials: Maren Rytter, PhD, Principal Investigator — Region Sjæland, Slagelse Hospital
Locations (1):
- Department of Paediatrics and Adolescent Medicine, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be made available to other researchers upon request

REFERENCES:
- [Background] Gavish R, Krause I, Goldberg L, Bilavsky E, Kadmon G, Livni G, Scheuerman O, Levinsky Y. A Drop in Number of Hospitalizations Among Children with Bacterial Infections During the COVID-19 Pandemic. Pediatr Infect Dis J. 2021 Jan;40(1):e39-e41. doi: 10.1097/INF.0000000000002963. PMID 33093429
- [Background] Kadambari S, Abo YN, Phuong LK, Osowicki J, Bryant PA. Decrease in Infection-related Hospital Admissions During COVID-19: Why Are Parents Avoiding the Doctor? Pediatr Infect Dis J. 2020 Nov;39(11):e385-e386. doi: 10.1097/INF.0000000000002870. No abstract available. PMID 32852351
- [Background] Kamrath C, Monkemoller K, Biester T, Rohrer TR, Warncke K, Hammersen J, Holl RW. Ketoacidosis in Children and Adolescents With Newly Diagnosed Type 1 Diabetes During the COVID-19 Pandemic in Germany. JAMA. 2020 Aug 25;324(8):801-804. doi: 10.1001/jama.2020.13445. PMID 32702751
- [Background] Foley DA, Yeoh DK, Minney-Smith CA, Martin AC, Mace AO, Sikazwe CT, Le H, Levy A, Moore HC, Blyth CC. The Interseasonal Resurgence of Respiratory Syncytial Virus in Australian Children Following the Reduction of Coronavirus Disease 2019-Related Public Health Measures. Clin Infect Dis. 2021 Nov 2;73(9):e2829-e2830. doi: 10.1093/cid/ciaa1906. No abstract available. PMID 33594407
- [Background] Polcwiartek LB, Polcwiartek C, Andersen MP, Ostergaard L, Broccia MD, Gislason GH, Kober L, Torp-Pedersen C, Schou M, Fosbol E, Kragholm K, Hagstrom S. Consequences of coronavirus disease-2019 (COVID-19) lockdown on infection-related hospitalizations among the pediatric population in Denmark. Eur J Pediatr. 2021 Jun;180(6):1955-1963. doi: 10.1007/s00431-021-03934-2. Epub 2021 Feb 8. PMID 33555426
- [Background] Nygaard U, Hartling UB, Nielsen J, Vestergaard LS, Dungu KHS, Nielsen JSA, Sellmer A, Matthesen AT, Kristensen K, Holm M. Hospital admissions and need for mechanical ventilation in children with respiratory syncytial virus before and during the COVID-19 pandemic: a Danish nationwide cohort study. Lancet Child Adolesc Health. 2023 Mar;7(3):171-179. doi: 10.1016/S2352-4642(22)00371-6. Epub 2023 Jan 9. PMID 36634692
- [Background] Fischer TK, Rungoe C, Jensen CS, Breindahl M, Jorgensen TR, Nielsen JP, Jensen L, Malon M, Braendholt V, Fisker N, Hjelt K. The burden of rotavirus disease in Denmark 2009-2010. Pediatr Infect Dis J. 2011 Jul;30(7):e126-9. doi: 10.1097/INF.0b013e3182145277. PMID 21386748